CLINICAL TRIAL: NCT03641638
Title: Correlation Between Different Levels of Thyroid Peroxidase Antibody and Postpartum Thyroiditis in Early Pregancy
Brief Title: Correlation Between Different Levels of Thyroid Peroxidase Antibody and Postpartum Thyroiditis in Early Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China National Nuclear Corporation 416 Hospital (Other)
Responsible Party: Principal Investigator, BO Ren, Attending physician, China National Nuclear Corporation 416 Hospital
Other Study IDs: CNNC416H
Record Dates: First submitted 2018-07-08; First posted 2018-08-22 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Postpartum Thyroiditis
Keywords: Postpartum thyroiditis; PPT; TPOAb
MeSH Terms: conditions — Postpartum Thyroiditis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Low level of TPOAb: normal thyroid function (FT3, FT4, TSH) before pregnancy, First pregnancy under 35 years old, early screening (1-12 weeks of pregnancy), initial screening of TPOAb positive, thyroid function: normal FT3 and FT4, TSH<4.78mIU/L，TPOAb at 34-102 IU/ml.
- Medium level of TPOAb: normal thyroid function (FT3, FT4, TSH) before pregnancy, First pregnancy under 35 years old, early screening (1-12 weeks of pregnancy), initial screening of TPOAb positive, thyroid function: normal FT3 and FT4, TSH<4.78mIU/L，TPOAb at 103-204 IU/ml.
- High level of TPOAb: normal thyroid function (FT3, FT4, TSH) before pregnancy, First pregnancy under 35 years old, early screening (1-12 weeks of pregnancy), initial screening of TPOAb positive, thyroid function: normal FT3 and FT4, TSH<4.78mIU/L，TPOAb >205IU/ml.
- Control group: normal thyroid function (FT3, FT4, TSH) before pregnancy, First pregnancy under 35 years old, early screening (1-12 weeks of pregnancy), initial screening of negative Thyroid antibody, thyroid function: normal FT3 and FT4, TSH<4.78mIU/L.

SUMMARY:
At present, attention to thyroid disease during pregnancy is increasing at home and abroad, but there is relatively little concern about postpartum thyroid disease, especially high incidence of postpartum thyroiditis (PPT). This observational study is to investigate the relationship between different levels of thyroid peroxidase antibody (TPOAb) and postpartum thyroiditis (PPT) in early pregnancy (1-12 weeks of pregnancy), and to explore whether PPT can be predicted by different TPOAb levels. According to the TPOAb level in early pregnancy, the postpartum of pregnant women was followed up, PPT was detected early, and intervention was performed according to thyroid dysfunction.

DETAILED DESCRIPTION:
First pregnant women who between the ages of 18 to 35 years old and normal thyroid function before pregnancy were selected. Recruit 300 pregnant women who early pregnancy (1-12 weeks of pregnancy) screening TPOAb positive and normal Free triiodothyronine (FT3), normal free thyroxine (FT4) ,Thyroid Stimulating Hormone (TSH) <4.78mIU / L as the observation group. They will be divided into low-level group (TPOAb at 34-102 IU/ml), medium-level group (TPOAb at 103-204 IU/ml), and high-level group (TPOAb>205) according to TPOAb. Recruit 100 pregnant women who early pregnancy (1-12 weeks of pregnancy) screening TPOAb negative and normal FT3, normal FT4,TSH <4.78mIU / L as the Control group.

Thyroid function (FT3, FT4, TSH) and TPOAb, thyroglobulin antibody(TgAb) ,thyroid hormone receptor antibody(TRAb) will be screened in the observation group and the control group at 3 months, 6 months, and 12 months after delivery. If the mother is diagnosed with postpartum thyroiditis (PPT), continue to screen for thyroid function (FT3, FT4, TSH) and thyroid antibodies (TPOAb, TRAb, TgAb) 18 months after delivery. The correlation between the early pregnancy TPOAb level and postpartum thyroiditis was analyzed between the observation group and the control group and the observation group. It was explored whether the occurrence of postpartum thyroiditis (PPT) can be predicted according to the TPOAb level in the first trimester. And targeted maternal effective follow-up and timely intervention to treat PPT provide important basis.

ELIGIBILITY:
Inclusion Criteria:

1. Observation group:

   * Pre-pregnancy tests for normal thyroid function (FT3, FT4, TSH)
   * First pregnancy between the ages of 18 to 35 years old
   * Early screening (1-12 weeks of pregnancy) initial screening TPOAb positive，thyroid function FT3, FT4 normal, TSH<4.78mIU/ L
2. Control group:

   * Pre-pregnancy tests for normal thyroid function (FT3, FT4, TSH) and antibodies
   * First pregnancy between the ages of 18 to 35 years old
   * Early pregnancy (1-12 weeks of pregnancy) initial screening negative thyroid-related antibody and thyroid function FT3, FT4 normal, TSH< 4.78 mIU/L.

Exclusion Criteria:

* Combined with other autoimmune diseases (such as systemic lupus erythematosus, etc.)
* Type 1 diabetes
* Gestational diabetes;
* Primary screening TRAb positive;
* Previous patients with Graves, subacute thyroiditis,chronic hepatitis
* Artificial pregnancy
* Suffering from liver and kidney dysfunction and other major diseases
* Have a history of adverse pregnancy
* Pregnant women with premature birth, miscarriage, intrauterine dysplasia and other unhealthy pregnancies withdrew from observation.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 300 pre-pregnancy tests for thyroid function (FT3, FT4, TSH) were normal, initial pregnancy under 30 years old, early screening (1-12 weeks of pregnancy), initial screening of TPOAb positive, thyroid function: normal FT3, FT4, TSH <4.78 mIU/L Females were observed and divided into low-level groups (TPOAb at 34-102 IU/ml), medium-level groups (TPOAb at 103-204 IU/ml), and high-level groups (TPOAb > 205 IU/ml) according to TPOAb.
  100 cases. 100 pre-pregnancy tests for thyroid function (FT3, FT4, TSH) and normal antibodies, first pregnancy under 30 years old, early pregnancy (1-12 weeks of pregnancy), initial screening for thyroid-related antibody negative and thyroid function: FT3, FT4 normal, TSH<4.78 Healthy women with mIU/L were the control group.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-08-31 (Estimated); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure the incidence rate of PPT in different TPOAb levels in early pregnancy. | 22 months
  The levels of TPOAb include:Low level of TPOAb(34-102 IU/ml),Medium level of TPOAb(103-204 IU/ml),High level of TPOAb(>205IU/m), TPOAb negative.

CONTACTS AND LOCATIONS:
Overall Officials: Ren Bo, Master, Principal Investigator — China National Nuclear Corporation 416 Hospital
Locations (1):
- China National Nuclear corporation 416 Hospital, Chengdu, Sichuan, China